CLINICAL TRIAL: NCT03581838
Title: Eating Behavior in Patients With Eosinophilic Esophagitis.
Brief Title: Eating With Eosinophilic Esophagitis (EoE)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Principal Investigator, Mayo Clinic
Other Study IDs: 18-002628
Record Dates: First submitted 2018-06-11; First posted 2018-07-10 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: EoE; Dysphagia
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acitve EoE: Observed eating session of Jimmy John's turkey or vegetarian sandwich with water among individuals who have EoE who have not been treated or have not achieved remission from treatment.
  Interventions: Behavioral: Observed eating session
- Remission EoE: Observed eating session of Jimmy John's turkey or vegetarian sandwich with water among individuals who have EoE who are have achieved remission from treatment.
  Interventions: Behavioral: Observed eating session
- Controls: Observed eating session of Jimmy John's turkey or vegetarian sandwich with water among individuals without EoE.
  Interventions: Behavioral: Observed eating session

INTERVENTIONS:
Behavioral: Observed eating session — Eating a Jimmy Johns turkey or vegetarian sandwich

SUMMARY:
Is there a difference in the eating process for patients with active Eosinophilic Esophagitis (EoE) and those with inactive disease?

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) patients develop adapted eating behaviors to prevent symptoms. These patients tend to cut their food small, chew extensively, take copious liquids with meals, and avoid foods that cause symptoms. No studies to date have directly evaluated these eating behaviors in patients with EoE with observation. Furthermore, none of the investigators' current metrics for patient symptom assessment visually evaluate the eating process nor are they compared before and after treatment. As a result, it is unclear if a patient's subjective perception of their eating difficulties and improvement matches with objective measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Patients suspected to have Eosinophilic Esophagitis
* Patients being treated for EoE with PPI or a steriod
* EoE patients that are in remission by having less than 22 on the EEsAI questionnaire
* Controls, patients that do not have EoE or other swallowing issues

Exclusion Criteria:

* Clinical evidence of infectious process potentially contributing to dysphagia (candidiasis, CMV,herpes)
* Other cause of dysphagia identified at endoscopy (reflux esophagitis, stricture, web, ring, achalasia, esophageal neoplasm)
* EoE patients that do not eat sandwiches or feel they could not eat a sandwich.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with EoE that are being seen at Mayo Clinic Esophageal Clinic will be approached. Controls will be individuals who do not have an EoE diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Observed eating session | 15-90 minutes
  number of bites of patient's with EoE and controls eating a Jimmy John's sandwich

SECONDARY OUTCOMES:
Food slowness during eating session | 15-90 minutes
  number of bites that felt stuck among patients with EoE and controls when eating a Jimmy John's sandwich
Water during eating session | 15-90 minutes
  amount of water drank of patients with EoE and controls eating a Jimmy John's sandiwch
Eosinophilic Esophagitis activity Index (EEsAI) questionnaire | 10-15 minutes
  The EEsAI Pro uses the VDQ is visual dysphagia question AMS is avoidance, modification, slow eating question . These two along with questions on frequency of, duration of, pain associated with dysphagia make up the PRO (patient reported outcomes). The PRO is a number (0-100) calculated from the answer to the questions. A PRO < 20 defines asymptomatic EoE.
Eosinophilic Esophagitis Quality of Life questionnaire | 10-15 minutes
  Higher score denote better quality of life. 0-4 as follows 4=not at all, 3=Slightly 2=moderately, 1=Quite a bit, 0= Extremely

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Alexander, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials